CLINICAL TRIAL: NCT04319133
Title: Effect Of Intermittent Fasting 5: 2 To Waist Circumference, Insulin Resistance And Oxidative Stress Marker In Obese Workers In Jakarta
Brief Title: Effect Of Intermittent Fasting To Metabolic And Oxidative Stress Marker
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Anni Rahmawati (Other)
Responsible Party: Sponsor-Investigator, Anni Rahmawati, Student, Indonesia University
Organization: Indonesia University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-02-0153
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Obesity
Keywords: obesity; intermittent fasting; insulin resistance; stress oxidative marker; waist circumference
MeSH Terms: conditions — Obesity; Intermittent Fasting; Insulin Resistance | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Intervention Model Description: Overall, this research will run for ± 10 weeks; 1 week of preparation, 8 weeks of intervention and 1 week of evaluation of the final results of the study.
  This research will involve an interview, physical examination and laboratory examination.
  This research is a clinical trial research with interventions in the form of fasting. There will be divided into two groups: the intervention group (fasting) and the control group (not fasting). The fasting group will fast every Monday and Thursday, while the fasting group consumes daily food as usual. Both groups will be given education about balanced nutrition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): Participants will ask to do 5:2 intermittent fasting (2 non-consecutive days a week) within 8 weeks
  Interventions: Behavioral: Fasting
- control (No Intervention): Participants will not doing fasting or intake restriction within 8 weeks

INTERVENTIONS:
Behavioral: Fasting — Doing fasting 2 days a week within 8 weeks
  Arms: intervention

SUMMARY:
The world prevalence of obesity in adult population in 2016 was 650 million while in Indonesia, it has increased from 14,8 percent to 21,8 percent in 2018. Obesity is an established risk factors for metabolic and non communicable- diseases. The purpose of this research was to assess the different effect on waist circumference, insulin resistance and oxidative stress marker between fasting (intervention) group and not fasting (control) group after 8 weeks 5:2 intermittent fasting (IF) among obese male workers.

DETAILED DESCRIPTION:
Intermittent fasting is eating pattern in that cycles between periods of fasting and eating. 5:2 intermittent fasting (IF) is a form of time-restricted fasting which no calories are consumed for at least 14 hours (for 4 am to 6 pm) will done in two non-consecutive days days per week, followed by ad libitum intake on the remaining days, with water restriction too.

Participants will be distributed to each group by simple randomization. This study will access the characteristic data, dietary intake and physical activity from the participants. Anthropometry and blood sample (for insulin resistance (HOMA-IR) and oxidative stress (malondialdehyde and catalase)) were taken at baseline and at the end of the study. Participants from each group will gets counseling at the second week of intervention and they will follow up to 8 weeks with control and evaluation form.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 30-59 years
* Has a BMI ≥ 25 kg/m^2
* Has a waist circumference of ≥ 90 cm
* Willingness to participate in the whole study by signing informed consent

Exclusion Criteria:

* Doing regular fasting (2 days a week) for 12 weeks before the study begins.
* In a certain diet at the moment
* Participants who are taking drugs that can affect blood sugar, insulin, and drugs (steroids, beta blockers, adrenergics), vitamins or herbal supplements and other drugs that affect oxidative stress.
* Participants suffering from obesity with complications such as impaired liver function, impaired kidney function, heart disease and type 2 diabetes mellitus are known through anamnesis and physical examination as well as fasting blood sugar checks.
* Participants that has a fever with temperatures> 37.5 ℃

Ages: 30 Years to 59 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — menstruating women will lose blood, so if they still asked to fast, it can endanger themselves because the nutrition is getting less
Enrollment: 62 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
insulin resistance | 8 weeks
  The pathological condition in which cells fail to respond normally to the hormone insulin. Assessed based on the HOMA-IR value
catalase level | 8 weeks
  Enzymatic antioxidant status of endogenous catalase in the blood, expressed in U/mg
plasma malondialdehyde level | 8 weeks
  the concentration of malondialdehyde (1,3-Propanedial) in the plasma as an oxidative stress marker measured by means of Will's method expressed in nmol/ml plasma unit
waist circumference | 8 weeks
  One way of anthropometry measurement to assess the visceral fat mass, so that it can evaluate the risk of metabolic disease. expressed in centimeter.

SECONDARY OUTCOMES:
mean caloric intake | 8 weeks
  the average amount of calories consumed daily by the participant which was determined from food diary and subsequent caloric contents calculation expressed in kilocalorie

CONTACTS AND LOCATIONS:
Overall Officials: Anni Rahmawati, postgraduate, Principal Investigator — Ilmu Gizi Fakultas Kedokteran Universitas Indonesia
Locations (1):
- PT DELAMITA BiILANO, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sutton EF, Beyl R, Early KS, Cefalu WT, Ravussin E, Peterson CM. Early Time-Restricted Feeding Improves Insulin Sensitivity, Blood Pressure, and Oxidative Stress Even without Weight Loss in Men with Prediabetes. Cell Metab. 2018 Jun 5;27(6):1212-1221.e3. doi: 10.1016/j.cmet.2018.04.010. Epub 2018 May 10. PMID 29754952
- [Result] Conley M, Le Fevre L, Haywood C, Proietto J. Is two days of intermittent energy restriction per week a feasible weight loss approach in obese males? A randomised pilot study. Nutr Diet. 2018 Feb;75(1):65-72. doi: 10.1111/1747-0080.12372. Epub 2017 Aug 9. PMID 28791787
- [Derived] Witjaksono F, Prafiantini E, Rahmawati A. Effect of intermittent fasting 5:2 on body composition and nutritional intake among employees with obesity in Jakarta: a randomized clinical trial. BMC Res Notes. 2022 Oct 12;15(1):323. doi: 10.1186/s13104-022-06209-7. PMID 36224641